CLINICAL TRIAL: NCT04048850
Title: Cohort Study of Hepatitis C Virus Treatment with Zepatier (Elbasvir/Grazoprevir) in Genotype 1 or 4 HCV Treatment-Naïve or Peginterferon/Ribavirin-Experienced Patients with Substance Use in Urban, Multidisciplinary Specialty Clinics
Brief Title: Zepatier in Patients with Substance Use
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Rodrigo Mauricio Burgos, Clinical Associate Professor, University of Illinois at Chicago
Other Study IDs: 2019-0478
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C; Hiv; Coinfection, HIV; Substance Use Disorders
Keywords: HCV; HIV-HCV coinfection; DAA; Elbasvir/grazoprevir
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; HIV Infections; Substance-Related Disorders | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients living with HCV +/- HIV: HCV monoinfected and human immunodeficiency virus (HIV)-HCV co-infected, HCV treatment-naïve or peginterferon/ribavirin-experienced patients with HCV genotype 1a, without baseline NS5A resistance, 1b, or 4 and substance use treated with elbasvir/grazoprevir 50-100 mg fixed-dose-combination, 1 tablet by mouth daily, for 12 weeks.
  Interventions: Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet [ZEPATIER]

INTERVENTIONS:
Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet [ZEPATIER] — Daily medication
  Other Names: Zepatier

SUMMARY:
The goal of this study is to assess hepatitis C virus (HCV) treatment with Zepatier (elbasvir/grazoprevir) in HCV monoinfected and human immunodeficiency virus (HIV)-HCV co-infected, HCV treatment-naïve or peginterferon/ribavirin-experienced patients with HCV genotype 1a, without baseline NS5A resistance, 1b, or 4 and substance use in urban, multidisciplinary specialty clinics.

DETAILED DESCRIPTION:
Previously, people who use substances and those without liver fibrosis or cirrhosis were excluded from receiving direct-acting antiviral (DAA) treatment due to Illinois Medicaid restrictions. These sobriety and staging restrictions were recently lifted. However, due to these previous stringent requirements for sobriety, many patients were not able to be treated for HCV. This created a data gap for real-world outcomes of HCV treatment in people who use substances. This study presents a unique opportunity to provide patients with hepatitis C treatment and obtain much needed data on the use of elbasvir/grazoprevir in patients with substance use and other underrepresented comorbidities. Additionally, this study will determine if our current standard of care for the treatment of HCV is effective for patients with substance use.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years of age or older)
* Chronic HCV (HCV antibody positive with detectable HCV-RNA)
* HCV genotypes 1a, without the presence of baseline NS5A resistance (specifically, polymorphisms at amino acid positions 28, 30, 31, or 93), 1b, or 4
* HCV treatment-naïve or peginterferon/ribavirin-experienced
* Managed by the UI Health Infectious Diseases Clinic or Liver Clinic
* Recent or current substance use (per self-report or electronic medical record (EMR) data within 90 days of the screening visit, with or without positive baseline urine toxicology), inclusive of one or more of the following: Opiate substitution therapy; Prescription medication misuse (including: opiates, sedatives, tranquilizers, hypnotics, and psychostimulants); Illicit substances; Injection drug use; Alcohol

Exclusion Criteria:

* Incarcerated
* Pregnant or breastfeeding
* Decompensated liver disease (Child-Pugh B or C)
* Albumin below 3 g/dL
* Platelet count below 75,000
* Unwilling to commit to treatment and/or monitoring
* Poor venous access inhibiting laboratory collection
* Any condition considered by the investigators to be a contraindication to study participation
* Hepatitis B virus (HBV) surface antigen (HBsAg) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The specific patient population to be studied is HCV monoinfected and HIV-HCV co-infected, HCV treatment-naïve or peginterferon/ribavirin-experienced patients of the UI Health Infectious Disease or Liver Clinic with HCV genotype 1a, without baseline NS5A resistance, 1b, or 4 and substance use treated with 12 weeks of elbasvir/grazoprevir therapy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
SVR - PP | 12 weeks after the end of therapy (SVR-12)
  Proportion of patients in the per-protocol (PP) population with sustained virologic response (SVR). PP: excludes non-treatment related discontinuations and patients lost to follow-up before SVR-12 laboratory test.

SECONDARY OUTCOMES:
SVR - stratified | 12 weeks after the end of therapy (SVR-12)
  PP SVR-12 stratified by pre-specified baseline characteristics:
  * HCV monoinfection
  * HIV-HCV co-infection
  * Cirrhosis
  * Positive baseline urine toxicology
  * Men who have sex with men (MSM)
  * Commercial sex work
  * Diagnosed concomitant psychiatric disorder(s)
  * Use of concomitant medication(s)
  * Specific substance(s) used
Drug-Drug interactions (DDIs) | From enrollment to treatment completion or termination, which ever comes first, for up to 36 weeks
  Interventions to prevent or remedy known or suspected DDIs between elbasvir/grazoprevir and concomitant prescription or over-the-counter medications, supplements, and substance of use
Adherence | During 12 weeks of treatment
  Self-reported adherence to elbasvir/grazoprevir, reported as number of missed doses and % missed doses of total doses
SVR - ITT | 12 weeks after the end of therapy (SVR-12)
  Proportion of patients in the intention-to-treat (ITT) population with SVR-12. ITT: all patients who received at least one dose of Zepatier (elbasvir/grazoprevir)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Mauricio Burgos, PharmD, Principal Investigator — University of Illinois at Chicago College of Pharmacy
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Illinois at Chicago Hospital and Health Sciences System — https://hospital.uillinois.edu/